CLINICAL TRIAL: NCT01223235
Title: A PILOT STUDY OF A POLYVALENT VACCINE-KLH CONJUGATE + OPT-821 GIVEN IN COMBINATION WITH BEVACIZUMAB IN PATIENTS WITH RECURRENT EPITHELIAL OVARIAN, FALLOPIAN TUBE, OR PRIMARY PERITONEAL CANCER WHO ARE IN SECOND OR GREATER COMPLETE OR PARTIAL CLINICAL REMISSION
Brief Title: Polyvalent Vaccine-KLH Conjugate + Opt-821 Given in Combination With Bevacizumab
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-099
Record Dates: First submitted 2010-10-14; First posted 2010-10-18 (Estimated); Results first posted 2018-05-14 (Actual); Last update posted 2018-06-12 (Actual); Status verified 2017-09

CONDITIONS: Fallopian Tubes Cancer; Ovarian Cancer; Peritoneal Cancer
Keywords: FALLOPIAN TUBE; OVARY; PERITONEUM; BEVACIZUMAB (AVASTIN); GLOBO H-KLH CONJUGATE; MUC-1 KLH; OPT-821; TF (C) - KLH; TN(C)-KLH; 10-099
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- bevacizumab & polyvalent vaccine-KLH conjugate + OPT-821 (Experimental): This is a single institution, open label, pilot study of bevacizumab and the polyvalent vaccine-KLH conjugate + OPT-821 in patients with recurrent epithelial ovarian, fallopian tube, or primary peritoneal cancer.
  Interventions: Biological: bevacizumab and the polyvalent vaccine-KLH conjugate + OPT-821

INTERVENTIONS:
Biological: bevacizumab and the polyvalent vaccine-KLH conjugate + OPT-821 — A maximum of 6 doses of the polyvalent-KLH vaccine and OPT-821 will be administered to each patient as per the schedule. Bevacizumab will be administered once every two weeks until week 11 and then once every three weeks according to the schedule. When the 6 vaccinations of the polyvalent-KLH vaccine +OPT821 are completed, patients may still continue to receive bevacizumab on the once every three week schedule.

SUMMARY:
The immune system of the body has the ability to fight and eliminate infections and cancers. Immune treatments, such as in this study, seek to teach the immune system to find and destroy cancer cells. The purpose of this study is to test whether it is safe to treat the cancer with a vaccine and another drug called bevacizumab (also known as Avastin).

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented epithelial carcinoma arising in the ovary, fallopian tube or peritoneum.
* Patients who have received cytoreductive surgery and chemotherapy with at least one platinum based chemotherapy regimen. Patients who received neoadjuvant chemotherapy are eligible.
* Patients with relapsed ovarian, fallopian tube or primary peritoneal cancer who have now completed chemotherapy and/or surgery for recurrent disease. Eligible patients are those who would be appropriate to enter a period of observation if standard management were considered.
* Patients who have asymptomatic residual measurable disease on CT scan or be in complete clinical remission. Patients may have an elevated CA-125. (Complete clinical remission is defined as serum CA-125 ≤ 35 IU/ml, negative physical examination and without objective evidence of disease by computed tomography (CT) of the abdomen and pelvis.)
* Adequate hematologic, coagulation, renal and hepatic function.
* ANC > = to 1,000 cells/mm3; platelets > or = 100,000 cells/mm3
* PT such that international normalized ratio (INR) is < 1.5 (or an in-range INR, usually between 2 and 3, if a patient is on a stable dose of therapeutic warfarin) Serum creatinine < or = to 1.5 mg/dl
* Bilirubin, SGOT, Alk Phos < 2.5x upper limit normal
* Urine protein : creatinine (UPC) ratio must be < 1 . If UPC ratio > 1, collection of 24-hour urine measurement of urine protein is recommended as part of the patient's medical management off-study.
* Karnofsky performance status > 70%
* Expected survival of at least 4 months
* Age ≥ 18 years. This protocol does not include children because the number of children with cancer is limited, and because a nationwide pediatric cancer research network already accesses the majority. Furthermore, the incidence of ovarian, fallopian tube, or peritoneal cancer in children is extremely infrequent.
* Patients who are ≥ 4 weeks from completion of prior cytotoxic chemotherapy. Prior bevacizumab and/or immunotherapy treatment are permitted

Exclusion Criteria:

* Inability to comply with study and/or follow-up procedures
* Current or recent (within 4 weeks of the first infusion of this study) participation in another experimental drug study.
* Active malignancy, other than superficial basal cell and superficial squamous (skin) cell, or carcinoma in situ of the cervix within last five years
* Patients must have undergone standard cytoreductive surgery as part of primary treatment to be eligible for this study and therefore are not of childbearing potential.Nursing mothers are excluded.
* Inadequately controlled hypertension (defined as systolic blood pressure >150 mmHg and/or diastolic blood pressure > 90 mmHg)
* Prior history of hypertensive crisis or hypertensive encephalopathy
* New York Heart Association (NYHA) Grade II or greater congestive heart failure (see Appendix C)
* History of myocardial infarction or unstable angina within 6 months prior to Day 1
* History of stroke or transient ischemic attack within 6 months prior to Day 1
* Known CNS disease, except for treated brain metastasis
* Treated brain metastases are defined as having no evidence of progression or hemorrhage after treatment and no ongoing requirement for dexamethasone, as ascertained by clinical examination and brain imaging (MRI or CT) during the screening period. Anticonvulsants (stable dose) are allowed. Treatment for brain metastases may include whole brain radiotherapy (WBRT), radiosurgery (RS; Gamma Knife, LINAC, or equivalent) or a combination as deemed appropriate by the treating physician. Patients with CNS metastases treated by neurosurgical resection or brain biopsy performed within 3 months prior to Day 1 will be excluded
* Significant vascular disease (e.g., aortic aneurysm, requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to Day 1
* History of hemoptysis (≥ 1/2 teaspoon of bright red blood per episode) within 1 month prior to Day 1
* Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation) or tumor involving major vessels.
* Major surgical procedure such as laparotomy, open biopsy, or significant traumatic injury within 28 days prior to Day 1 or anticipation of need for major surgical procedure during the course of the study
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to Day 1
* History of abdominal fistula or gastrointestinal perforation within 6 months prior to Day
* Patients with clinical symptoms or signs of GI obstruction who require parenteral hydration, parenteral nutrition, or tube feeding
* Patients with evidence of abdominal free air not explained by paracentesis or recent surgical procedure
* Serious, non-healing wound, active ulcer, or untreated bone fracture
* Known hypersensitivity to any component of bevacizumab
* Allergy to seafood
* Active autoimmune disease (i.e. rheumatoid arthritis, ulcerative colitis etc); or immune deficiency (HIV, hypogammaglobulinemia); or known active infections with Hepatitis B or Hepatitis C; or those receiving immunosuppressive drugs (such as chronic systemic corticosteroids or cyclosporin, etc); or those receiving chronic antiinflammatory drugs (intermittent use of anti-inflammatory drugs is permitted).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-10; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Sabbatini, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Kahn RM, Ragupathi G, Zhou QC, Iasonos A, Kravetz S, Hensley ML, Konner JA, Makker V, Tew WP, Aghajanian C, Sabbatini PJ, O'Cearbhaill RE. Long-term outcomes of patients with recurrent ovarian cancer treated with a polyvalent vaccine with bevacizumab combination. Cancer Immunol Immunother. 2023 Jan;72(1):183-191. doi: 10.1007/s00262-022-03225-1. Epub 2022 Jul 2. PMID 35779095
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bevacizumab & Polyvalent Vaccine-KLH Conjugate + OPT-821
Started | 22
Completed | 21
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Bevacizumab & Polyvalent Vaccine-KLH Conjugate + OPT-821
Number analyzed (Participants) | 22
Age, Continuous [Median (Full Range); unit: years] | 56 [49 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 22
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Toxicities evaluated by CTCAE version 4.0
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab & Polyvalent Vaccine-KLH Conjugate + OPT-821
Number analyzed (Participants) | 21
Participants | 21

2. Secondary Outcome: Percentage of Participants Who Met the Immunogenicity Criteria (>/=3 Antigens) of the Vaccine
Description: when given in the presence of bevacizumab
  Patients must have IgM titer >1:80, or a fourfold increase in prevailing antibody titer if present at baseline. Twenty-one patients would be accrued, and if >8 of 21 patients should meet these criteria for three or more antigens based on the immune response criteria, the study would be considered positive.
Time Frame: 1 year
Measure: Number; unit: % of participants
Arm/Group | Bevacizumab & Polyvalent Vaccine-KLH Conjugate + OPT-821
Number analyzed (Participants) | 21
% of participants | 68

3. Secondary Outcome: Progression-free Survival as Assessed By Multiplex Biomarker Panel of Angiogenesis Markers
Description: Progression is defined as at least a 20% increase in the sum of diameters of target lesions. The sum must also demonstrate an absolute increase of at least 5mm.
Time Frame: Up to 24 months
Measure: Median (95% Confidence Interval); unit: months (Progression Free Survival)
Arm/Group | Bevacizumab & Polyvalent Vaccine-KLH Conjugate + OPT-821
Number analyzed (Participants) | 21
months (Progression Free Survival) | 13 [10 to 20]

ADVERSE EVENTS:
Time Frame: Until time to treatment failure, up to 20 months.
Arm/Group | Bevacizumab & Polyvalent Vaccine-KLH Conjugate + OPT-821
All-Cause Mortality (participants affected / at risk) | 18/21
Serious Adverse Events (participants affected / at risk) | 5/21
Other Adverse Events (participants affected / at risk) | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab & Polyvalent Vaccine-KLH Conjugate + OPT-821 (N=21)
Acute Kidney Injury (Renal and urinary disorders) | 1
Chest pain - cardiac (Cardiac disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Fatigue (General disorders) | 1
Fever (General disorders) | 2
Injection site reaction (General disorders) | 1
Urinary tract obstruction (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab & Polyvalent Vaccine-KLH Conjugate + OPT-821 (N=21)
Injection site reaction (General disorders) | 3
Headache (Nervous system disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Fever (General disorders) | 3
White blood cell decreased (Investigations) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 3
Nausea (Gastrointestinal disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Blood bilirubin increased (Investigations) | 1
Diarrhea (Gastrointestinal disorders) | 1
Serum amylase increased (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-06-12): https://cdn.clinicaltrials.gov/large-docs/35/NCT01223235/Prot_SAP_000.pdf